CLINICAL TRIAL: NCT04507568
Title: The Person-centered Evolution of Radiotherapy Services in Ontario (PERSON) Study
Brief Title: The Person-centered Evolution of Radiotherapy Services in Ontario Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-5111
Record Dates: First submitted 2020-07-29; First posted 2020-08-11 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Quality of Life
Keywords: Radiation Therapy; Patient Experience; Anxiety Levels
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Person-Centered Model-of-Care (Experimental): Patients randomized to the person-centered model-of-care will have a 30 minute education session with a radiation therapist in addition to the standard of care, radiation therapy procedures.
  Interventions: Other: Quality of Life Questionnaires
- Standard Model-of-Care (Other): Patients randomized to the standard model of care will be treated as per standard of care.
  Interventions: Other: Quality of Life Questionnaires

INTERVENTIONS:
Other: Quality of Life Questionnaires — Quality of Life questionnaires will be administered to both arms at baseline, and at the first and last day of treatment.

SUMMARY:
This is a single center, prospective, investigator initiated, randomized controlled study of patients with breast cancer who will be receiving radiation therapy as per SOC. Patients will be randomized in either the person-centered model-of-care versus the standard model of care.

Patients randomized to the person-centered model-of-care will have a 30 minute education session with a radiation therapist in addition to RT SOC procedures. Patients randomized to the standard model of care will be treated as per SOC. Questionnaires will be administered to both arms at baseline, and at the first and last day of treatment. In addition to the main study, patients will have the option to participate in a semi-structured one on one interview upon completion of their radiotherapy course.

DETAILED DESCRIPTION:
Radiation therapy plays an integral role in the definitive treatment of breast cancer by reducing the risk of locoregional recurrence and improving patient outcomes. Despite the availability of supportive care services, many patients have unmet needs which may lead to unexpected negative outcomes. Anxiety can affect patients' ability to cope, interfere with treatment and self-manage their own care. Strategies to improve cancer care include patient navigators or case managers, early interventions and self-management of side effects to reduce treatment-related toxicities. Therefore, minimizing distress from treatment and engaging patients by personalizing care according to their unique needs will optimize use of supportive care services and improve clinical outcomes.

A Cochrane review demonstrated that information and supportive care sessions delivered by non-physician healthcare providers improves both emotional wellbeing and quality of life in breast cancer patients. A prospective randomized, Australian study by Halkett et al. demonstrated that an education intervention delivered one-on-one by Radiation Therapists effectively reduces breast cancer patients' psychological distress and improves preparedness for treatment. This highlights the importance of early and accessible education resources where patients experience direct access to the radiation therapy team.

Further research is required to investigate the efficacy of person-centered model on patient experiences and relevant clinical outcomes. Specifically, it is expected this model will reduce patient anxiety, improve preparedness for radiation therapy through education, and improve patient self-management of radiation-toxicities. The proposed study focuses on patients with breast cancer because of the experience in testing the model on this group and their relatively uniform treatment at all Ontario cancer centres, which will facilitate translation of this model in the future. A randomized controlled study will determine the efficacy of the person-centered model versus standard care, and generate high-quality evidence in an unbiased setting that was not possible in the prior clinical pilot phases.

Personalizing patient experiences in radiotherapy, coupled with improvements in treatment quality and supportive care, may improve clinical outcomes including toxicity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Diagnosis of non-metastatic breast cancer
* Intended to receive radiation therapy to the breast/chest-wall and regional lymph nodes
* Ability to communicate in English without assistance of another person
* Ability to provide informed consent

Exclusion Criteria:

* Commenced any radiation therapy-specific procedures (e.g. education, CT-simulation, etc.)
* Received a previous course of radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Patient Anxiety Levels | Up to 5 weeks.
  Hospital Anxiety and Depression Scale (HADS) questionnaire

SECONDARY OUTCOMES:
Patient-reported self-efficacy | Up to 5 weeks.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Self Efficacy Survey
Patient-reported engagement level | Up to 5 weeks.
  Patient Health Engagement (PHE) survey
Patient-reported experience | Up to 5 weeks.
  EORTC satisfaction with cancer care core (EORTC PATSAT-C33) questionnaire
Patient-reported experience | Up to 5 weeks.
  Specific complementary outpatient module (EORTC OUT-PATSAT7) questionnaire
Patient-reported preparedness for radiation therapy | Up to 5 weeks.
  Cancer Treatment Survey (CaTS)

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada